CLINICAL TRIAL: NCT01051700
Title: A Two-part Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Repeat Oral Doses of Pazopanib in Healthy Adult Subjects
Brief Title: A Safety Study in Healthy Volunteers to Evaluate Safety, How Fast the Drug is Absorbed, and the Side Effects of the Drug in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 113555
Record Dates: First submitted 2010-01-07; First posted 2010-01-18 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Macular Degeneration
Keywords: repeat-dose; pharmacokinetics; choroidal neovascularization; safety; GW786034; tolerability; age-related macular degeneration; stem cell growth factor; pazopanib; platelet derived growth factor; vascular endothelial growth factor
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — pazopanib

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 5 mg (Experimental): GW786034
  Interventions: Drug: GW786034
- 10 mg (Experimental): GW786034
  Interventions: Drug: GW786034
- 20 mg (Experimental): GW786034
  Interventions: Drug: GW786034
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GW786034 — Investigational product
  Other Names: pazopanib
  Arms: 10 mg; 20 mg; 5 mg
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is to evaluate the safety, absorption rate and side effects associated with the study drug. Healthy volunteers will be given a single dose of the drug in Part 1. Subjects will be dosed at the same time at several different sites. In Part 2 of the study elderly volunteers will participate in a 14 day repeat dose session receiving either study drug or a placebo (sugar pill). Data from at least 7 days of safety will be reviewed from the first set of volunteers before increasing the doses for the next set. All results will be used for planning the next study.

DETAILED DESCRIPTION:
The purpose of this study is to characterize more fully the safety, tolerability and pharmacokinetics of single and repeat oral doses of pazopanib at lower doses than those previously studied. The first part of the study is designed as an open-label, non-randomized, single session, parallel-group, sequential dose-rising to investigate pharmacokinetics of single oral doses in healthy adult subjects. In the second part of the study, healthy elderly subjects will participate in one 14 day repeat-dose session, randomized to receive either pazopanib or placebo. Dose escalation within Part 2, is based upon emerging safety and PK data from each preceding repeat dosing cohort from at least 7 days of safety data as well as emerging safety and PK data from single dose. The elderly population chosen for the second part of the study will more closely reflect the target population for the AMD indication. The results from the current study will assist in the dose selection of the subsequently planned study in patients with AMD.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin less than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* For the first part of the study male or female greater than or equal to 18 years of age and for the second part male or female greater than or equal to 50 years of age at the time of signing the informed consent.
* A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea. In questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) or values consistent with local laboratory recommended value is confirmatory.
* Body weight greater than or equal to 50 kg for men and greater than or equal to 45 kg for women within the BMI range 19-30 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Single QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.
* Best-corrected visual acuity better than 20/80 (Snellen equivalent) in both eyes in Part 2 only.

Exclusion Criteria:

* History of clinically relevant impaired endocrine, thyroid, hepatic, respiratory or renal function, uncontrolled hypertension, diabetes mellitus, coronary heart disease, or psychotic mental illness.
* History of any clotting disorder, including predisposition to hypercoagulation or any previous thromboembolic event.
* Elevations in blood pressure, based on criteria provided in Section 7.2.3. OR Subjects with a blood pressure >140/90 mmHg, at screening.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as: For US sites: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prohibited medications as described in Section 9.2.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Any prior intraocular surgery, excluding cataract surgery (Part 2 only)
* Any prior eye surgery within three months to first dose of study medication (Part 2 only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-01-12 (Actual); Primary Completion 2010-05-27 (Actual); Study Completion 2010-05-27 (Actual)

PRIMARY OUTCOMES:
Clinical safety data from AE reporting, clinical observations, physical exam findings, cardiac monitoring, vital signs, clinical laboratory tests, Pharmacokinetics, general ophthalmic examination and best-corrected visual acuity will be summarized. | 4 months

SECONDARY OUTCOMES:
Pharmacokinetic parameters: AUC vs time curve after single dose; AUC vs time curve, trough plasma pazopanib concentration, accumulation ratio, and apparent terminal half-life after repeat dose will be analyzed, as data permit | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Tacoma, Washington

REFERENCES:
- [Derived] McLaughlin MM, Paglione MG, Slakter J, Tolentino M, Ye L, Xu CF, Suttle AB, Kim RY. Initial exploration of oral pazopanib in healthy participants and patients with age-related macular degeneration. JAMA Ophthalmol. 2013 Dec;131(12):1595-601. doi: 10.1001/jamaophthalmol.2013.5002. PMID 24113783
- See also: Results for study 113555 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/113555?search=study&study_ids=113555#rs